CLINICAL TRIAL: NCT03076554
Title: A Pilot Study to Investigate the Safety and Clinical Activity of Avelumab (MSB0010718C) in Thymoma and Thymic Carcinoma After Progression on Platinum-Based Chemotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170066; 17-C-0066
Record Dates: First submitted 2017-03-09; First posted 2017-03-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09-22

CONDITIONS: Thymoma; Thymic Carcinoma
Keywords: Programmed Death 1 (PD-1); Immune Checkpoint Blockade
MeSH Terms: conditions — Thymoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — avelumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 Avelumab (Experimental): Avelumab will be administered at a dose of 10 mg/kg intravenously once every two weeks until disease progression or development of intolerable adverse events.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Avelumab will be administered at a dose of 10 mg/kg intravenously once every two weeks until disease progression or development of intolerable adverse events.

SUMMARY:
Background:

Thymoma and thymic carcinoma are cancers originating in the thymus gland. Platinum-based chemotherapy is standard treatment for them. But not uncommonly, the disease returns and people need more treatment to keep the cancer from growing. The drug Avelumab could help the immune system fight cancer.

Objective:

To test if avelumab is safe and well-tolerated, and is effective in treating relapsed or refractory thymoma and thymic carcinoma.

Eligibility:

People ages 18 and older with thymoma or thymic carcinoma that has returned or progressed after platinum-containing chemotherapy

Design:

Participants will be screened with:

* Blood, urine, and heart tests
* Scan: They lie in a machine that takes pictures of the body.
* Physical exam
* Medical history
* Biopsy: a needle removes a piece of tumor. Samples can be from a previous procedure, although it is desirable to undergo a new biopsy.

Participants will have treatment in 2-week cycles. They will continue until the side effects are not tolerable or their disease gets worse. Visits at the following time points are required per protocol. Patients who respond to treatment or have durable stability after at least 12 months of therapy may undergo a dose de-escalation regimen to continue on therapy.

* Every 2 weeks: Participants will get avelumab by infusion in a vein (IV). They will get diphenhydramine (benadryl) and acetaminophen (tylenol) by mouth or IV before receiving avelumab to decrease the chances of developing a reaction to avelumab. They will have blood, urine, and heart tests periodically.
* Cycles 4 and 7, then every 6 weeks: Scans will be performed to look for shrinkage or growth of tumor.
* Cycle 4: Participants will be offered a chance to undergo a biopsy.
* 2-4 weeks after stopping treatment: Blood, urine, and heart tests will be performed. Participants might undergo a scan.
* 10 weeks after stopping treatment: Blood, urine, and heart tests.
* About 6 months after stopping treatment, then every 3 months: Participants will have scans andcan allow genetic testing on their blood and tissue samples.

DETAILED DESCRIPTION:
Background

Platinum-based chemotherapy is the standard of care for advanced unresectable thymic epithelial tumors (TETs). However more than half of these patients experience disease recurrence and require second-line therapy. There are no approved drugs for treatment of recurrent thymoma and thymic carcinoma and new therapeutic options are needed for patients who have disease progression on or after platinum-containing therapy. The clinical activity of checkpoint blockade targeting programmed death 1 (PD-1) and its ligand (PD-L1) has been demonstrated against various tumor types. We have demonstrated the ability of avelumab to induce major responses in patients with advanced thymoma in a phase I dose escalation study. Further investigation of avelumab in patients with TETs is needed to define the clinical activity and safety of immune checkpoint blockade in patients with TETs.

Primary Objectives

To determine the safety and tolerability of avelumab in participants with relapsed or refractory thymoma and thymic carcinoma.

To determine the objective response rate (ORR) to avelumab in participants with relapsed or refractory thymoma and thymic carcinoma.

Eligibility

Participants with histologically confirmed, unresectable thymoma or thymic carcinoma who have previously been treated with at least one platinum-containing chemotherapy regimen with progressive disease prior to study entry

Prior treatment with immune checkpoint inhibitors is permitted if the reason for discontinuation was not disease progression or life-threatening adverse events (laboratory abnormalities alone with prior therapy will not exclude participants from this trial)

Measurable disease by RECIST 1.1 criteria

Adequate renal, hepatic and hematopoietic function

No major surgery, radiotherapy, chemotherapy or biologic therapy within 28 days of avelumab

No prior thymic tumor-associated autoimmune disease with the exception of pure red cell aplasia and vitiligo.

Design

This will be a single-arm, pilot study to determine the clinical activity and safety of treatment with avelumab in participants with relapsed or refractory thymoma and thymic carcinoma.

Avelumab will be administered at a dose of 10 mg/kg intravenously once every two weeks until disease progression or development of intolerable adverse events. The two week period will constitute one cycle.

Per the study team s discretion, participants who respond to treatment or have durable stability after at least 12 months of therapy may undergo a dose de-escalation regimen to continue on therapy.

Toxicity will be assessed every cycle by CTCAE version 5.0.

Tumor response will be assessed after completion of every third cycle (6 weeks) using RECIST criteria, version 1.1.

When possible, a tumor biopsy will be conducted pre-treatment and on C4D43 to evaluate treatment-related, intra-tumoral changes.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically confirmed thymoma or thymic carcinoma by the pathology department/CCR/NCI.
* Participants must have had at least one prior line of platinum-based chemotherapy or participant must have refused cytotoxic chemotherapy. Progressive disease must be documented prior to study entry and participants must have advanced, unresectable disease that is not amenable to surgical resection.
* Prior treatment of PD-1 or PD-L1-directed immune checkpoint blockade is permitted if treatment was not discontinued due to disease progression or lifethreatening adverse events per the investigators discretion (laboratory abnormalities alone with prior therapy will not exclude participants from this trial).
* Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1.
* Individuals aged greater than or equal to 18 years

  -- Because no dosing or adverse event data are currently available on the use of Avelumab in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status less than or equal to 1.
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count: greater than or equal to 1,500/mm^3 OR greater than or equal to 1.5 x 10^9/L
  * platelets greater than or equal to 100,000/mm^3 OR greater than or equal to 100 x 10^9/L
  * hemoglobin greater than or equal to 9g/dL (may have been transfused)
  * total bilirubin less than or equal to 1.5 x the upper limit of normal range(ULN)
  * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 x ULN OR less than or equal to 5 x ULN for participants with documented metastatic disease to the liver
  * creatinine clearance greater than or equal to 30 mL/min according to the Cockcroft Gault formula (or local institutional standard method)
* Highly effective contraception for all individuals if the risk of conception exists. (Note: The effects of the study drug on the developing human fetus are unknown. Thus, individuals of childbearing potential and those able to father a child must agree to use highly effective contraception, defined as 2 barrier methods, or 1 barrier method with a spermicide, an intrauterine device or use of oral female

contraceptive. Effective contraception must be used 30 days prior to first study drug administration, for the duration of trial participation, and at least 30 days after last avelumab treatment administration if the risk of conception exists. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this trial, the treating physician should be informed immediately.)

* Pregnancy test: negative serum or urine pregnancy test at screening for women of childbearing potential.
* Ability of individual to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Concurrent treatment with a non-permitted drug
* Concurrent anticancer treatment within 28 days before the start of trial treatment (e.g., cytoreductive therapy, radiotherapy [with the exception of palliative bone directed radiotherapy], immune therapy, or cytokine therapy except for erythropoietin); major surgery within 28 days before the start of trial treatment (excluding prior diagnostic biopsy); concurrent systemic therapy with immunosuppressive agents within 28 days before the start of trial treatment; use of hormonal agents for the treatment of thymic cancer within 7 days before the start of trial treatment; or use of any investigational drug within 28 days before the start of trial treatment.

  --Note: Individuals receiving bisphosphonate or denosumab are eligible provided treatment was initiated at least 14 days before the first dose of avelumab.
* History of previous malignant disease within the last 2 years with the following exceptions: basal or squamous cell carcinoma of the skin, cervical carcinoma in situ, ductal carcinoma in situ of the breast, papillary or follicular thyroid carcinoma, and non-muscle invasive bladder cancer.
* Active autoimmune disease that might deteriorate when receiving an immune-stimulatory agent. Participants with diabetes type 1, vitiligo, psoriasis, pure red cell aplasia, Good s syndrome or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible. Anti-acetylcholine receptor antibodies will be checked during screening. Participants will be ineligible if results are positive, even if there is no clinical history of autoimmune disease.
* Participants with symptomatic brain metastases will be excluded from trial secondary to poor prognosis. However, participants who have had treatment for their brain metastasis and whose brain disease has remained stable for 3 months without steroid therapy may be enrolled.
* Active infection requiring systemic therapy or significant acute or chronic infections including, among others:

  * Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive).
  * Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
* Prior organ transplantation including allogenic stem-cell transplantation.
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5 Grade greater than or equal to 3).
* Persisting toxicity related to prior therapy (NCI CTCAE v5Grade > 1) however, alopecia, sensory neuropathy Grade less than or equal to 2, or other Grade less than or equal to 2 not constituting a safety risk based on investigator s judgment are acceptable.
* Pregnancy or lactation period. Note: a negative pregnancy test is required for individuals of childbearing potential. Individuals who are postmenopausal (age-related amenorrhea greater than or equal to 12 consecutive months or follicle-stimulating hormone (FSH) > 40 milli international units per milliliter [mIU/ml]), or who had undergone hysterectomy or bilateral oophorectomy are exempt from pregnancy testing. If necessary to confirm postmenopausal status a FSH level will be included at screening.
* Pregnant individuals are excluded from this study because Avelumab is in the class of agents known as antineoplastics/monoclonal antibodies with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in

nursing infants secondary to treatment of the mother with Avelumab, breastfeeding should be discontinued if the mother is treated with Avelumab.

* Known alcohol or drug abuse.
* Clinically significant (i.e. active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (>= New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* All other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participants inappropriate for entry into this study.
* Any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Legal incapacity or limited legal capacity.
* Non-oncology vaccine therapies for prevention of infectious disease (e.g. seasonal flu vaccine, human papilloma virus vaccine) within 4 weeks of study drug administration with the exception of vaccinations against COVID-19. Vaccination while on study is also prohibited except for administration of inactivated vaccines (e.g. inactivated influenza vaccines) and vaccinations against COVID-19.
* HIV-positive TET participants are ineligible because of the risk of developing opportunistic infections after treatment with an immune checkpoint inhibitor. Prior cases of disseminated herpes virus and fungal infections have been documented in this patient population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of Avelumab based on NCI-CTCAE v4.0 | End of every cycle
  Toxicity profile based on NCI-CTCAE v4.0
Objective Response Rate (ORR) based on RECIST 1.1 criteria | Every other cycle
  Objective response rate; i.e., the number of participants with complete response + the number with partial response confirmed via RECIST 1.1

SECONDARY OUTCOMES:
Immune-related progression-free survival (irPFS) | Date of progression
  Immune-related progression-free survival
Overall Survival (OS) | Date of death
  Overall survival
Duration of Response | Date of progression
  Time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Katsuya Y, Fujita Y, Horinouchi H, Ohe Y, Watanabe S, Tsuta K. Immunohistochemical status of PD-L1 in thymoma and thymic carcinoma. Lung Cancer. 2015 May;88(2):154-9. doi: 10.1016/j.lungcan.2015.03.003. Epub 2015 Mar 10. PMID 25799277
- [Background] Padda SK, Riess JW, Schwartz EJ, Tian L, Kohrt HE, Neal JW, West RB, Wakelee HA. Diffuse high intensity PD-L1 staining in thymic epithelial tumors. J Thorac Oncol. 2015 Mar;10(3):500-8. doi: 10.1097/JTO.0000000000000429. PMID 25402569
- [Derived] Remon J, Girard N, Novello S, de Castro J, Bigay-Game L, Bernabe R, Greillier L, Mosquera J, Cousin S, Juan O, Sampayo M, Besse B. PECATI: A Multicentric, Open-Label, Single-Arm Phase II Study to Evaluate the Efficacy and Safety of Pembrolizumab and Lenvatinib in Pretreated B3-Thymoma and Thymic Carcinoma Patients. Clin Lung Cancer. 2022 May;23(3):e243-e246. doi: 10.1016/j.cllc.2021.07.008. Epub 2021 Jul 20. PMID 34393061
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0066.html